CLINICAL TRIAL: NCT02227342
Title: A Prospective, Single Center, Open Label Trial of Fecal Microbiota Transplantation (FMT) in the Management of Active Ulcerative Colitis
Brief Title: Fecal Microbiota Transplantation (FMT) in the Management of Active Ulcerative Colitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Dina Kao, Associate Professor, University of Alberta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 47056
Record Dates: First submitted 2014-07-22; First posted 2014-08-28 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fecal Microbiota Transplantation (Experimental): serial Fecal Microbiota Transplantation
  Interventions: Biological: Fecal Microbiota Transplant

INTERVENTIONS:
Biological: Fecal Microbiota Transplant — serial FMT

SUMMARY:
Manipulation of the intestinal microbiota through FMT is a potential therapeutic target for IBD patients. Studies are now required to determine if repeated FMT can overcome the apparent immune response to FMT thereby maintaining sustained clinical improvement and remission. Prior to a large randomized controlled trial of FMT in UC we will carry out a feasibility study to determine if serial FMTs can sustain a clinical response and maintain stability of transplanted microbiota.

DETAILED DESCRIPTION:
same as above

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 and < 65 years
2. Diagnosis of UC for > 3 months but < 5 years prior to screening as determined by the investigators
3. Those with mild to moderate UC
4. Those who have failed maintenance therapy with stable doses of 5-ASA, azathioprine or 6 mercaptopurine (6-MP) for > 3 months
5. Where applicable, those who are taking the following medications must be at a stable dose defined as:

   i) 5-ASA must be at a stable dose for 2 weeks ii) Prednisone up to 20 mg/d must be at a stable dose for 2 weeks iii) Budesonide up to 6 mg/d must be at a stable dose for 2 weeks iv) Azathioprine or 6-MP must be at a stable dose for > 8 weeks
6. ability to provide informed consent
7. evidence of active inflammation

Exclusion Criteria:

1. Those whose disease is limited to the rectum (ie. proctitis)
2. Those with colectomy or diverting ileostomy
3. Those who are pregnancy or plan to be pregnant during the trial
4. Those who are breastfeeding or plan to breast feed during the trial
5. Those who are on or have previously failed a biological agent
6. Those with an active infection requiring antibiotic therapy
7. Those with positive stool cultures for known pathogens such as E coli, Salmonella, Shigella, Yersinia, Campylobacter, and Clostridium difficile toxin within 2 weeks of enrollment
8. Those with positive CMV on colonic tissue biopsy within 2 weeks of screening
9. Those with allergy to ciprofloxacin and metronidazole
10. Those with colonic mucosal dysplasia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Mayo score reduction | 12 and 32 weeks
  Patients with at least 3 point reduction in partial Mayo scoring index at week 12 and at week 32 in the extension phase.

CONTACTS AND LOCATIONS:
Overall Officials: Dina Kao, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada